CLINICAL TRIAL: NCT03634592
Title: A Prospective Registry of Atrial Fibrillation Ablation Using the Prediction of Lesion Depth Technology
Brief Title: AF Ablation With the Ablation Index
Status: Completed | Type: Observational
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Sponsor
Other Study IDs: AF0718NR
Record Dates: First submitted 2018-08-02; First posted 2018-08-16 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Catheter ablation — Radiofrequency catheter pulmonary vein isolation

SUMMARY:
This is an observational multicenter registry of atrial fibrillation catheter ablation performed using the ablation index technology.

DETAILED DESCRIPTION:
This is an observational multicenter registry of atrial fibrillation catheter ablation performed using the ablation index technology, which has been introduced as a tool predicting ablation lesion depth. The index incorporates the following characteristics of radiofrequency point-by-point ablation: radiofrequency energy power, contact force, duration of ablation. Since the ablation index is calculated for every individual operator depending on his(her) personal skills, there is no a strict indication on the safe and effective range of the index. This registry aims to evaluate ablation index values used in different centers by different operators. Prospective information on arrhythmia recurrence rate and type, characteristics of redo ablations, characteristics of reconduction ablated areas will be gathered.

ELIGIBILITY:
Inclusion Criteria:

* indications for catheter ablation of atrial fibrillation;
* signed informed consent

Exclusion Criteria:

* Presence of contraindications to AF ablation

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (both males and females aged 18-79 years) with indications to atrial fibrillation ablation undergoing radiofrequency catheter pulmonary vein isolation
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Freedom from atrial fibrillation | 1 year
  Number of participants with no evidence of atrial tachyarrhythmia longer than 30 s in duration at 12 months after ablation, as detected by regular ECG monitoring according to centres' established practices (Holter monitoring every 3 months, implantable loop recorder, cardiac rhythm management device interrogation, other regular ECG screening). Data will be collected using a web-based system with electronic case report forms.

SECONDARY OUTCOMES:
Acute complications | 30 days
  Number of participants with adverse events that are related to treatment (i.e. cardiac tamponade, periprocedural stroke, pulmonary vein stenosis, esophageal damage, etc) whithin 30 days after ablation. Data will be collected using a web-based system with electronic case report forms.
Procedure time | 180 minutes
  Duration of the total ablation procedure and fluoroscopy needed to complete pulmonary vein isolation, expressed in minutes.
Fluoroscopy time | 24 hours
  Fluoroscopy duration within the procedure
Electrical reconduction | 2 years
  Number of participats with electrical reconduction into pulmonary veins as assessed during repeat procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal State Budgetary Institution "V. A. Almazov Federal North-West Medical Research Centre" of the Ministry of Health of the Russian Federation, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided